CLINICAL TRIAL: NCT01345734
Title: Liraglutide Effectiveness and Safety Data From Routine Clinical Practice in Philippines Study. A Multicentre, Open Label, Observational, Non-interventional Study to Evaluate the Safety and Effectiveness of Liraglutide in Subjects With Type 2 Diabetes Mellitus in Philippines
Brief Title: Non-Interventional Study on Safety of Liraglutide in Subjects With Type 2 Diabetes
Acronym: Lead-Ph
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-3932; U1111-1119-8803 (Other: WHO)
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Liraglutide will be prescribed and titrated by the treating physician and will be self-administered by the subject s.c. (under the skin) once daily. Study participants being treated with GLP-1 (Glucagon-Like Peptide 1)agonists or DDP-4-inhibitors (Dipeptidyl-peptidase 4 ) should stop treatment when initiating liraglutide treatment.

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the safety profile of liraglutide under normal conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus, including newly-diagnosed subjects or those already receiving other anti-diabetic medications including GLP-1 analogues other than Liraglutide, who require treatment with liraglutide according to the clinical judgment of their treating physician
* Subjects who are capable of giving study-specific signed informed consent before any collection of information

Exclusion Criteria:

* Subjects with type 1 diabetes
* Subjects who are or have previously been on liraglutide
* Subjects who are participating in another clinical trial
* Subjects with a hypersensitivity to liraglutide or to any of the excipients (Disodium phosphate dihydrate, propylene glycol, phenol, water for injections)
* Subjects who are pregnant, breast feeding or have the intention of becoming pregnant within the following 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult subjects with type 2 diabetes, including newly-diagnosed subjects or those already receiving other anti-diabetic medications including GLP-1 analogues other than liraglutide.
Sampling Method: Non-Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2013-07-26 (Actual); Study Completion 2013-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence of serious adverse drug reactions (SADRs) | Week 0, week 26

SECONDARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) | Week 0, week 26
Incidence of serious adverse events (SAEs) | Week 0, week 26
Frequency of hypoglycaemic episodes | Week 0, week 26
Change in HbA1c (glycosylated haemoglobin)" | Week 0, week 26

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Manila, Philippines

REFERENCES:
- [Result] Jimeno C, Kho S, de Los Santos GK, Buena-Bobis N, Villa M. The Multicenter, Open-Label, Observational LEAD-Ph Study: Real-World Safety and Effectiveness of Liraglutide in Filipino Participants with Type 2 Diabetes. J ASEAN Fed Endocr Soc. 2018;33(2):114-123. doi: 10.15605/jafes.033.02.02. Epub 2018 Oct 9. PMID 33442116
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com